CLINICAL TRIAL: NCT01859715
Title: Hepatic Cytochrome Drug Interactions in Emergency Department Patients
Brief Title: Emergency Department (ED) Drug Interaction in Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-1692
Record Dates: First submitted 2013-05-01; First posted 2013-05-22 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Drug Interactions
Keywords: Drug Interactions; CYP2D6; opioid efficacy; pain; nausea
MeSH Terms: conditions — Pain; Nausea | interventions — Oxycodone; Hydrocodone; acetaminophen, hydrocodone drug combination; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxycodone group (Active Comparator): Subjects given either oxycodone 5mg by ED provider decision or by triage nurse randomization.
  Interventions: Drug: Oxycodone
- Nausea-observational group (Active Comparator): Patients given ondansetron 4mg by ED provider decision or by triage nurse. This is an observational cohort only.
  Interventions: Drug: Ondansetron
- Hydrocodone/Acetaminophen group (Active Comparator): Subjects given hydrocodone/acetaminophen 5mg/500mg by ED provider decision or by triage nurse randomization.
  Interventions: Drug: Hydrocodone

INTERVENTIONS:
Drug: Oxycodone — Subjects given oxycodone 5mg by ED provider decision or by triage nurse randomization.
  Other Names: Oxycodone, oxycontin
  Arms: Oxycodone group
Drug: Hydrocodone — Subjects given hydrocodone/acetaminophen 5mg/500mg by ED provider decision or by triage nurse randomization.
  Other Names: Vicodin
  Arms: Hydrocodone/Acetaminophen group
Drug: Ondansetron — Subjects given ondansetron 4mg for reported nausea or vomiting. Treatment determined either by triage nursing protocol or by provider discretion. Observational intervention only.
  Other Names: Zofran
  Arms: Nausea-observational group

SUMMARY:
This study examines how hepatic cytochrome CYP2D6 drug interactions affects the efficacy of oxycodone, hydrocodone, and ondansetron in Emergency Department (ED) patients.

DETAILED DESCRIPTION:
Patients with pain and/or nausea are enrolled in the Emergency Department (ED). They are given either oxycodone, hydrocodone, or ondansetron at the discretion of the Emergency Department (ED) provider or the triage nurse by triage protocol. Detailed prescription, over the counter, herbal, supplement, and illicit drug ingestion histories are taken from the patient or their health care proxy. Serial visual analogue scales are captured prior to study drug administration then between 30 and 90 minutes following drug administration.

ELIGIBILITY:
Inclusion Criteria:

* self-reported pain or nausea identified by the initial nursing assessment

Exclusion Criteria:

* unable to speak English,
* < 18 y.o.,
* previously diagnosed with chronic pain or cyclic vomiting

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Monte, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated in the University of Colorado Hospital ED. A convenience sample sample of ED patients were enrolled between June 2012 to January 2013. Subjects were included if they had self-reported pain or nausea identified during the initial nursing assessment. The previous 2 day medication history was obtained during their visit.
Pre-assignment Details: 201/502 consented patients did not receive the study medication. The remaining 301 patients were allocated to either one of the opioid treatment groups or the nausea observational group based on what study medication they were prescribed and if they were able to complete serial visual analog scales for pain and nausea.
Groups:
- Oxycodone Group: Subjects given oxycodone 5mg by ED provider decision or by triage nurse randomization.
- Nausea-observational Group: Patients given ondansetron 4mg for reported nausea or vomiting by ED provider decision or by triage nurse. This is an observational cohort only.
Period: Overall Study
Arm/Group | Oxycodone Group | Hydrocodone/Acetaminophen Group | Nausea-observational Group
Started | 141 | 91 | 116
Completed | 125 | 83 | 93
Not Completed | 16 | 8 | 23
Not completed — No 2nd VAS | 16 | 8 | 23

BASELINE CHARACTERISTICS:
Groups:
- Hydrocodone/Acetaminophen Group: Subjects given hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
- Nausea-observational Group: Patients given ondansetron for reported nausea or vomiting by ED provider decision or by triage nurse. This is an observational cohort only.
- Total: Total of all reporting groups
Arm/Group | Oxycodone Group | Hydrocodone/Acetaminophen Group | Nausea-observational Group | Total
Number analyzed (Participants) | 141 | 91 | 116 | 348
Age, Continuous [Mean (Full Range); unit: years] | 40 [18 to 86] | 38 [18 to 84] | 34 [18 to 85] | 40 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 56 | 83 | 218
  Male | 62 | 35 | 33 | 130
Number of CYP2D6 drugs taken [Median (Full Range); unit: CYP2D6 drug] | 1 [0 to 6] | 1 [0 to 5] | 1 [0 to 6] | 1 [0 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Difference in Clinically Significant Visual Analogue Scale for Pain and Nausea Change Between CYP2D6 Users and Non-users
Description: Clinically significant visual analogue scale (VAS; a measure of adult pain and nausea on a scale of 1-100 millimeters for increasing symptoms of pain and nausea) for patients who were administered either oxycodone, hydrocodone/acetaminophen, or ondansetron in the ED. Clinically significant change was defined as 13mm change on the VAS from baseline (when first VAS was completed) to 90 minutes following drug administration in the ED.
Time Frame: Baseline and 90 minutes
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- Oxycodone Group: Subjects given oxycodone 5mg mg by ED provider decision or by triage nurse randomization.
- Hydrocodone/Acetaminophen Group: Subjects given or hydrocodone/acetaminophen 5mg/500mg by ED provider decision or by triage nurse randomization.
Arm/Group | Oxycodone Group | Hydrocodone/Acetaminophen Group | Nausea-observational Group
Number analyzed (Participants) | 125 | 83 | 93
millimeters | 7.4 [-0.8 to 15.6] | 10.9 [0.8 to 21.1] | -14.0 [-23.6 to -4.4]

2. Secondary Outcome: Adverse Drug Events
Description: Determine all possible adverse drug events that occurred after the study drugs were administered.
Time Frame: Duration of ED stay, <24 hours. (up to 24 hours)
Measure: Number; unit: participants
Arm/Group | Oxycodone Group | Hydrocodone/Acetaminophen Group | Nausea-observational Group
Number analyzed (Participants) | 125 | 83 | 93
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Oxycodone Group; Hydrocodone/Acetaminophen Group: Subjects given either oxycodone 5mg or hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
  Oxycodone: Subjects given either oxycodone 5mg or hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
  Hydrocodone: Subjects given either oxycodone 5mg or hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
- Nausea-observational Group: Patients given ondansetron by ED provider decision or by triage nurse. This is an observational cohort only.
  Oxycodone: Subjects given either oxycodone 5mg or hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
  Hydrocodone: Subjects given either oxycodone 5mg or hydrocodone/acetaminophen 5mg/500 mg by ED provider decision or by triage nurse randomization.
  Ondansetron: Subjects given ondansetron for reported nausea or vomiting. Treatment determined either by triage nursing protocol or by provider discretion. Observational intervention only.
Arm/Group | Oxycodone Group | Hydrocodone/Acetaminophen Group | Nausea-observational Group
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/91 | 0/116
Other Adverse Events (participants affected / at risk) | 0/141 | 0/91 | 0/116

LIMITATIONS AND CAVEATS:
These data are limited by the nature of self-reported medication ingestion histories and self-reported effectiveness measures for opioid pain medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes